CLINICAL TRIAL: NCT03322813
Title: A Study to Evaluate the Safety and Feasibility of Exablate Model 4000 Type-2 to Temporarily Mediate Blood-Brain Barrier Disruption (BBBD) in Patients With Suspected Infiltrating Glioma in the Setting of Planned Surgical Interventions
Brief Title: ExAblate Blood Brain Barrier Disruption (BBBD) for Planned Surgery in Suspected Infiltrating Glioma
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study temporarily suspended until priorities are reassessed
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT004
Record Dates: First submitted 2017-10-19; First posted 2017-10-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Glioma
Keywords: Glioblastoma; Blood Brain Barrier; BBB; ExAblate; Blood Brain Barrier Disruption; Infiltrating glioma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ExAblate 4000 - Type 2 (Experimental): ExAblate BBBD
  Interventions: Device: ExAblate 4000 - Type 2

INTERVENTIONS:
Device: ExAblate 4000 - Type 2 — Using ExAblate Model 4000 Type-2 to temporarily disrupt the blood brain barrier in non-enhancing suspected infiltrating glioma undergoing resection
  Other Names: ExAblate BBBD

SUMMARY:
This study is designed to assess the safety and feasibility of using the ExAblate, Type 2 to temporarily disrupt the blood brain barrier in non-enhancing suspected infiltrating glioma. The ExAblate Model 4000 Type-2 is intended for use as a tool to disrupt the BBB.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, non-randomized, open-label feasibility study to evaluate the safety of focal BBBD using the ExAblate® 4000 Type 2 system. Up to 15 subjects with suspected infiltrating glioma who are scheduled to undergo brain tumor resection may be recruited for the study. Only patients that have a non-enhancing tumor components in a non-eloquent region of the planned standard-of-care resection volume will be eligible. Up to 4 centers may participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female between 21-85 years of age
2. Able and willing to give informed consent
3. Subjects with suspected infiltrating glioma on pre-operative brain imaging scans including non-enhancing MRI tumor components in non-eloquent regions that are within the planned surgical resection volume
4. Surgical area targeted for ExAblate treatment (i.e. prescribed Region of Treatment) ≤30 cm3; planned surgical resection volume may exceed the targeted treatment volume
5. Karnofsky Performance Score 70-100
6. Able to communicate sensations during the ExAblate® BBBD procedure

Exclusion Criteria:

1. MRI or clinical findings of:

   * Active or chronic infection(s) or inflammatory processes
   * Acute or chronic hemorrhages, specifically any lobar microbleeds, and no siderosis, amyloid angiopathy, or macrohemorrhages
   * Intracranial thrombosis, vascular malformation, cerebral aneurysm or vasculitis
   * Evidence of tumor-related calcification, cyst, or hemorrhage
   * Midline shift of >10mm or evidence of subfalcine, uncal, or tonsillar herniation on pre-operative imaging
2. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
3. Clips, shunts, or any metallic implanted objects in the skull or the brain or the presence of unknown MR unsafe devices anywhere within the body
4. Significant cardiac disease or unstable hemodynamic status
5. Uncontrolled hypertension (systolic > 150 and diastolic BP > 100 on medication)
6. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk of hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
7. History of a liver disease, bleeding disorder, coagulopathy or a history of spontaneous hemorrhage
8. Abnormal coagulation profile (Platelets < 100,000), PT (>14) or PTT (>36), and INR > 1.3
9. Lacunar lesions or evidence of increased risk of bleeding
10. Known cerebral or systemic vasculopathy
11. Significant depression and at potential risk of suicide
12. Known sensitivity/allergy to gadolinium, or other intravascular contrast agents
13. Active seizures despite medication treatment (defined as >1 seizure per month) which could be worsened by disruption of the blood brain barrier
14. Evidence of worsening neurological function
15. Dexamethasone dose ≥ 24mg daily or equivalent steroid dose
16. History of drug or alcohol disorder which have a higher risk for seizures, infection and/or poor executive functioning
17. Positive HIV status, which can lead to increased entry of HIV into the brain parenchyma leading to HIV encephalitis
18. Potential blood-borne infections which can lead to increased entry to brain parenchyma leading to meningitis or brain abscess
19. Any contraindications to MRI scanning, including:

    * Large subjects not fitting comfortably into the scanner
    * Difficulty lying supine and still for up to 3 hours in the MRI unit or claustrophobia
20. Untreated, uncontrolled sleep apnea
21. Impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
22. Respiratory: chronic pulmonary disorders e.g. severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area, patients with a history of drug allergies, asthma or hay fever, and multiple allergies where the benefit/risk of administering Definity® is considered unfavorable by the study physicians in relation to the product labeling for Definity
23. Currently in a clinical trial involving an investigational product or non-approved use of a drug or device

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Device and procedure related adverse events | At the time of the ExAblate MRgFUS procedure
  The number and severity of device and BBBD procedure related adverse events will be evaluated.

SECONDARY OUTCOMES:
Feasibility of BBB disruption | At the time of the ExAblate MRgFUS procedure and 24 hours post-procedure
  The extent and reversibility of BBB opening will be determined by the degree of contrast enhancement seen on post-procedure MRI with contrast agent

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Woodworth, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Medical System, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Anastasiadis P, Gandhi D, Guo Y, Ahmed AK, Bentzen SM, Arvanitis C, Woodworth GF. Localized blood-brain barrier opening in infiltrating gliomas with MRI-guided acoustic emissions-controlled focused ultrasound. Proc Natl Acad Sci U S A. 2021 Sep 14;118(37):e2103280118. doi: 10.1073/pnas.2103280118. PMID 34504017